CLINICAL TRIAL: NCT00833105
Title: Rehabilitation of the Upper Extremity With Enhanced Proprioceptive Feedback Following Incomplete Spinal Cord Injury (SCI)
Brief Title: Rehabilitation of the Upper Extremity With Enhanced Proprioceptive Feedback Following Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Paul J. Cordo, Study Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4649; NCT00437515 (obsolete NCT alias)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury; Tetraplegia; Paresis; Plegia
Keywords: Incomplete Spinal Cord Injury; Rehabilitation; Upper Extremity; AMES device; Incomplete SCI; Quadriplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paresis; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMES treatment (Experimental): The subject will receive 25 treatment sessions, conducted 2-3 times per week on the AMES device. Each session will consist of testing followed by 30 minutes of wrist and finger rehabilitation using the AMES device.
  Interventions: Device: AMES treatment

INTERVENTIONS:
Device: AMES treatment — The AMES device rotates the fingers-thumb or the wrist in the flexion-extension directions over a range of 30 degrees while vibrators stimulate the tendons attached to muscles that are lengthened by the thumb-finger or hand movement. A treatment consists of 20 minutes of fingers-thumb movement, followed by 10 minutes of wrist movement. The subject's task is to assist the motion of the device.

SUMMARY:
The purpose of this study is to determine if tetraplegic individuals with incomplete spinal cord injury (SCI) who remain unable to move their arms normally 1 year after their SCIs are able to sense and move the affected arm(s) better after 10-13 weeks of treatment with a new robotic therapy device.

The hypothesis is that using the AMES device on the arm(s) of chronic tetraplegic subjects with incomplete SCI will result in improved strength, sensation, and functional movement in treated limb(s).

DETAILED DESCRIPTION:
Traumatic spinal cord injury (SCI) affects over 200,000 people in the USA, with several thousand new injuries each year. Most recovery, following SCI, occurs in the six months following surgery. Further recovery after 12 months is unusual.

In this study 13 subjects, more than 1 year post injury, were enrolled to test the safety and efficacy of a new type of robotic therapy device known as the AMES device. The aim of this Phase I/II study is to investigate the use of assisted movement and enhanced sensation (AMES) technology in hand rehabilitation of incomplete SCI subjects.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI with tetraplegia.
* Male or female.
* 18-65 yrs old.
* At least 1 yr post-SCI.
* Tolerate sitting upright at for at least one hour.
* Able to perceive direction of passive joint(s) motion of the upper extremity(ies) to be treated 70% or more of the times tested.
* Motor grade >1 in the wrist extensors, finger flexors and finger abductors (the 3 muscles related to hand movements in the ASIA scale) in the upper extremity tested.
* Cognitively and behaviorally capable of complying with the regimen.

Exclusion Criteria:

* Fracture of the treated limb resulting in loss of range of motion
* Concomitant TBI or stroke (Patients who sustained mild head injury during the trauma with no evidence of structural abnormalities on brain images will qualify for the study)
* DVT of the treated extremity
* Peripheral nerve injury of the treated extremity
* Osteo- or rheumatoid-arthritis limiting range of motion
* Contractures equal to or greater than 50% of the normal ROM
* Skin condition not tolerant of device
* Progressive neurodegenerative disorder
* Botox treatment of the treated extremity in the prior 5 month
* Chronic ITB therapy
* Uncontrolled seizure disorder
* Uncontrolled high blood pressure/angina
* Pain in affected limb or exercise intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Cordo, Ph.D, Principal Investigator — Oregon Health and Science University; Deborah Backus, PhD, PT, Principal Investigator — Shepherd Center, Atlanta GA
Locations (2):
- United States (2):
  - Shepherd Center, Atlanta, Georgia
  - Oregon Health and Science University, Portland, Oregon

REFERENCES:
- [Result] Cordo P, Lutsep H, Cordo L, Wright WG, Cacciatore T, Skoss R. Assisted movement with enhanced sensation (AMES): coupling motor and sensory to remediate motor deficits in chronic stroke patients. Neurorehabil Neural Repair. 2009 Jan;23(1):67-77. doi: 10.1177/1545968308317437. Epub 2008 Jul 21. PMID 18645190

RESULTS

PARTICIPANT FLOW:
Groups:
- AMES Treatment: The subject will receive 25 treatment sessions, conducted 2-3 times per week on the AMES device. Each session will consist of testing followed by 30 minutes of wrist and finger rehabilitation using the AMES device.
  AMES treatment: The AMES device rotates the fingers-thumb or the wrist in the flexion-extension directions over a range of 30 degrees while vibrators stimulate the tendons attached to muscles lengthened by the finger or wrist movements. A treatment consists of 20 minutes of fingers-thumb movement, followed by 10 minutes of wrist movement. The subject's task is to assist the motion of the device.
Period: Overall Study
Arm/Group | AMES Treatment
Started | 13
Completed | 10
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Enrolled 13 subjects. Three subjects dropped out. Of the remaining 10 subjects, 15 limbs were tested, both limbs in 5 of the subjects.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Age at time of injury [Mean (Standard Deviation); unit: years] | 41.5 (14.1)
ASIA Motor Key Muscles [Mean (Standard Deviation); unit: units on a scale] — Measures the level of impairment of key muscles controlling the upper limb, including: elbow flexors (spinal level C5), wrist extensors (spinal level C6), elbow extensors (spinal level C7), finger flexors (spinal level C8), and finger abductors (spinal level T1). The scale range is 0 (total paralysis) to 5 (normal active movement), but also includes a scale category "NT," which indicates that muscle group was not testable. Total score is the sum of the scores from all 5 spinal levels ranging from 0-25. A higher score means less upper limb impairment.
  units on a scale | 15.6 (3.6)
Time since injury [Mean (Standard Deviation); unit: years] | 3.5 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Grasp Release Test
Description: The task involves picking up, transporting, and placing six objects (i.e., peg, paperweight, fork, block, can, and videotape). Movement of each of the 6 objects is scored based on the number of times the participant can move the object in 30 seconds, with a minimum score of zero if no objects are successfully moved. A cumulative score is based on the sum of all completed movements for all 6 objects.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Error); unit: Objects moved
Units Other Than Participants: Arms
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Arms) | 15
Objects moved
  Pre-training | 58.5 (37.9)
  Post-training | 72.0 (40.0)
  3 Month Follow-up | 77.5 (44.9)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p < 0.025, Mixed Models Analysis; Random subject effect

2. Secondary Outcome: ASIA Motor Key Muscles
Description: ISNCSCI Assessment of motor function (upper limb only). Scores on a scale ranging from 0 (i.e., total paralysis) - 5 (i.e., full range of motion) for each of 5 upper limb muscle groups. Total score represents the overall level of the upper limb impairment and represents the sum of the 5 scores from the 5 upper limb muscle groups. Accordingly, the total score has a range of 0-25, with 0 representing a completely paralyzed upper limb and 25 representing a normally functioning upper limb.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
units on a scale
  Pre-training | 15.3 (3.9)
  Post-training | 14.6 (4.4)
  3 Month Follow-up | 16.1 (4.7)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p = 0.299, Mixed Models Analysis; Random subject effect

3. Secondary Outcome: ASIA (ISNCSCI) Sensory/Key Sensory Points/ Light-Touch
Description: Measures the subject's sensory perception, with eyes closed, of a light touch by the tester on 9 key sensory points of the hand, arm, shoulder and neck. Sensation at each key point is rated as a number on a scale from 0 (no feeling) to 2 (normal feeling), with a score of 1 representing partly diminished feeling. The overall sensation of the upper limb and nearby areas is represented as the sum of all 9 individual key point scores and, therefore, has an overall range of 0-18, with higher scores representing better sensation.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
units on a scale
  Pre-training | 14.1 (3.3)
  Post-training | 13.8 (3.3)
  3 Month Follow-up | 14.5 (3.1)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p = 0.459, Mixed Models Analysis; Random subject effect

4. Secondary Outcome: ASIA (ISNCSCI) Sensory/Key Sensory Points/Pin-Prick
Description: Measures the subject's sensory perception, with eyes closed, of a light prick of a safety pin produced by the tester on 9 key sensory points of the hand, arm, shoulder and neck. Sensation at each key point is rated as a number on a scale from 0 (no feeling) to 2 (normal feeling), with a score of 1 representing partly diminished feeling. The overall sensation of the upper limb and nearby areas is represented as the sum of all 9 individual key point scores and, therefore, has an overall range of 0-18, with higher scores representing better sensation.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
units on a scale
  Pre-training | 10.5 (5.4)
  Post-training | 11.3 (5.3)
  3 Month Follow-up | 11.1 (4.6)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p = 0.343, Mixed Models Analysis; Random subject effect

5. Secondary Outcome: Van Lieshout Hand Function Test for Tetraplegia- Short Version
Description: Measures the functional movement in the upper limb of people with cervical spinal cord injury. The short version of this test includes a total of 10 different functional tasks to be performed by the subject with the upper limb. For example, one task is to reach and pick up a filled Coke bottle, set it down, and then replace it in its original position. Each task is scored on a scale of 0-5, 0 representing inability to perform the task and 5 representing normal movement. A single, total score is calculated as the sum of the scores on the 10 tasks, and therefore, has an overall range of 0-50, with higher scores representing better performance.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
units on a scale
  Pre-training | 27.2 (11.8)
  Post-training | 27.3 (11.1)
  3 Month Follow-up | 27.4 (12.6)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p = 0.951, Mixed Models Analysis; Random subject effects

6. Secondary Outcome: Modified Ashworth Scale
Description: Measurement of joint stiffness (tone/spasticity). Score is based on sum of MAS value for 4 muscle groups: (1) Wrist/finger flexors, (2) Wrist/finger extensors, (3) elbow flexors, and (4) elbow extensors. Each muscle group and direction is score on a scale of 0 (no increase in muscle tone) to 5 (rigid), with a score of 2 used instead of 1+. A single overall score representing the sum of all 4 muscle groups and directions is used and has a range of 0-20 with higher scores representing more severe impairment.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
units on a scale
  Pre-training | 5.3 (3.4)
  Post-training | 4.4 (3.2)
  3 Month Follow-up | 4.2 (3.3)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p = 0.371, Mixed Models Analysis; Random subject effect

7. Secondary Outcome: Capabilities of Upper Extremity Instrument
Description: Subjective questionnaire of participants' self-perceptions of upper limb function that contains 17 questions relating to the use of the right upper limb, the same 17 relating to the use of the lower upper limb, plus two additional questions relating to bimanual function. Responses to each item of the questionnaire has a range of 1 (i.e., "totally limited") to 7 (i.e., "not at all limited"). A total cumulative score used for the study is based on the sum of the responses to all 34 questions (i.e., 16 right arm, 16 left arm, 2 both arms), and therefore has a cumulative score range of 32 - 224, with higher scores indicating more function.
Time Frame: Prior to training (baseline), after 25 training sessions (about 8 weeks), 3 months post-training
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
units on a scale
  Pre-training | 58.2 (23.0)
  Post-training | 64.1 (24.6)
  3 Month Follow-up | 63.8 (25.8)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p = 0.164, Mixed Models Analysis; Random subject effect

8. Secondary Outcome: Strength Test - Thumb/Finger Extension
Description: Maximum strength of thumb-and-fingers in extension.
  Pre-training score is average of a total of 3 scores, including 1 score from each of the first 3 days of training. Post-training score is average of a total of 3 scores, including 1 score from each of the last 3 days of training.
Time Frame: Prior to training (baseline), after each of 25 training sessions (about 3 times/week)
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: Newton*meters
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
Newton*meters
  Pre-training | 0.43 (0.43)
  Post-training | 0.65 (0.65)
Statistical Analysis 1: Comparison: AMES Treatment; Pre-training score is average of a total of 9 efforts, including 3 efforts from the first 3 days of training. Post-training score is average of a total of 9 efforts, including 3 efforts from the last 3 days of training; Test type: Superiority or Other; p < 0.01, Wilcoxon Signed-Rank; No multiple comparison procedure

9. Secondary Outcome: Strength Test - Thumb/Fingers Flexion
Description: Maximum strength of Thumb/fingers in Flexion
  Pre-training score is average of a total of 9 efforts, including 3 efforts from the first 3 days of training. Post-training score is average of a total of 9 efforts, including 3 efforts from the last 3 days of training.
Time Frame: Prior to training (baseline), after each of 25 training sessions (about 3 times/week)
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: Newton*meters
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
Newton*meters
  Pre-training | 2.10 (1.75)
  Post-training | 2.87 (2.94)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p < 0.05, Wilcoxon Signed Rank Test — No multiple comparison procedure performed

10. Secondary Outcome: Strength Test - Wrist Extension
Description: Maximum wrist strength in extension
  Pre-training score is average of a total of 9 efforts, including 3 efforts from the first 3 days of training. Post-training score is average of a total of 9 efforts, including 3 efforts from the last 3 days of training.
Time Frame: Prior to training (baseline), after each of 25 training sessions (about 3 times/week)
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: Newton*meters
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
Newton*meters
  Pre-training | 2.27 (1.50)
  Post-training | 3.51 (2.02)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test — No multiple comparison procedure

11. Secondary Outcome: Strength Test - Wrist Flexion
Description: Maximum strength in flexion direction
  Pre-training score is average of a total of 9 efforts, including 3 efforts from the first 3 days of training. Post-training score is average of a total of 9 efforts, including 3 efforts from the last 3 days of training.
Time Frame: Prior to training (baseline), after each of 25 training sessions (about 3 times/week)
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: Newton*meters
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
Newton*meters
  Pre-training | 5.41 (3.31)
  Post-training | 7.95 (4.98)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p < 0.005, Wilcoxon Signed Rank Test — No multiple comparison adjustment

12. Secondary Outcome: Active Motion Test - Fingers/Thumb
Description: Tracking task for the thumb and finger, i.e., opening and closing the hand. The participant tracks a target box on a video screen by actively moving the thumb and fingers, first in the opening direction, then closing, and finally opeining again. The participant's thumb-and-finger position is represented on the video screen by a vertical line that he/she attempts to keep in the the target box. Performance on this task is scored as the amount of time, in seconds, that the participant keeps the line in the target box. The maximum total score in this test is 60 seconds. The "Pre-training Score" is the average score obtained during the first 3 days of training, and the Post-training Score" is average score obtained during the last 3 days of training.
Time Frame: Prior to training (baseline), after each of 25 training sessions (about 3 times/week)
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
Seconds
  Pre-training | 6.95 (5.98)
  Post-training | 10.63 (7.20)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — No multiple comparison adjustment

13. Secondary Outcome: Active Motion Test - Wrist
Description: Tracking task for the wrist, i.e., flexing (i.e., pull with the front of the hand) and extending (i.e., pushing with the back of the hand). The participant tracks a target box on a video screen by actively moving the hand at the wrist, first in the extension direction, then flexion, and finally extension again. The participant's wrist position is represented on the video screen by a vertical line that he/she attempts to keep in the the target box. Performance on this task is scored as the amount of time, in seconds, that the participant keeps the line in the target box. The maximum total score in this test is 60 seconds. The "Pre-training Score" is the average score obtained during the first 3 days of training, and the Post-training Score" is average score obtained during the last 3 days of training.
Time Frame: Prior to training (baseline), after each of 25 training sessions (about 3 times/week)
Population: Analysis population is "arms." Three subjects dropped out. Five of the remaining subjects were tested for both arms.
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Upper Limbs
Arm/Group | AMES Treatment
Number analyzed (Participants) | 10
Number analyzed (Upper Limbs) | 15
Seconds
  Pre-training | 18.50 (11.27)
  Post-training | 26.62 (11.77)
Statistical Analysis 1: Comparison: AMES Treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — No multiple comparisons adjustment

ADVERSE EVENTS:
Time Frame: Time of enrollment until completing the 3-month follow-up evaluation (i.e., 5-6 months)
Arm/Group | AMES Treatment
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMES Treatment (N=13)
Liver disease requiring hospitalization (Hepatobiliary disorders) | 1 (1)
Suicide (Psychiatric disorders) | 1 (1) — Presumed due to depression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMES Treatment (N=13)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Reduction in tenodesis (Musculoskeletal and connective tissue disorders) | 1 (1) — Strength gain in finger flexors reduced ability to use tenodesis
Bleeding (Blood and lymphatic system disorders) | 1 (1) — Subject accidentally pricked on ear lobe during sensory testing producing 1 drop of blood.
Skin abrasion (Skin and subcutaneous tissue disorders) | 2 (2) — Abrasion from vibrator probe
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Tripped over dog and fractured shoulder
Muscular soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — After first training session

LIMITATIONS AND CAVEATS:
1. Not a controlled study.
2. Zone of partial preservation not fully characterized.
3. Changes in somatosensation were not quantified.
4. Five participants were trained for both ULs, so training of first UL may have affected second UL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No